CLINICAL TRIAL: NCT01125202
Title: Intervention to Reduce Dietary Sodium in Hemodialysis
Acronym: BalanceWise-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Iowa (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mary Ann Sevick, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08040361; R01NR010135 (NIH)
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Renal Dialysis
Keywords: Intervention studies; Computers, handheld; Randomized controlled trial; Sodium, dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCT-based behavioral intervention (Experimental): Intervention participants continue to receive routine dialysis care, as well as a 16 week dietary counseling intervention based on Social Cognitive Theory. Dietary counseling is paired with Personal Digital Assistant-based dietary self-monitoring.
  Interventions: Behavioral: SCT-based behavioral intervention
- Attention control (Active Comparator): Attention control participants continue to receive routine dialysis care. Attention control participants view 5 computerized educational programs PowerPoint slides) that summarize the various elements of the HD diet. The 5 modules evenly over the 4-month study period.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: SCT-based behavioral intervention — Intervention group continues to receive routine dialysis care. The intervention duration is 16 weeks. Intervention contacts are 2x/week for weeks 0-8, weekly for weeks 9-12, and every other week for weeks 13-16. Personal digital assistant dietary records are use to provide targeted counseling and engaged the participant in problem solving around dietary issues.
  Arms: SCT-based behavioral intervention
Behavioral: Attention Control — Attention control participants continue to receive routine dialysis care. Attention control participants view 5 computerized educational programs PowerPoint slides) that summarize the various elements of the HD diet. The 5 modules evenly over the 4-month study period.
  Arms: Attention control

SUMMARY:
The purpose of this study is to test, in a randomized clinical trial of 200 hemodialysis patients, a behavioral intervention to reduce dietary sodium intake. The investigators will assess the impact on weight gain between dialysis treatments, blood pressures, symptoms, and health-related quality of life. The primary study hypotheses are that participants will gain less weight in between dialysis treatments, and that dietary recalls will demonstrate reduced consumption of dietary sodium.

DETAILED DESCRIPTION:
Cardiovascular disease is the single most common cause of death in hemodialysis (HD) patients. Most HD patients have left ventricular hypertrophy(LVH), a significant predictor of death in this population. LVH is related to extracellular volume expansion and hypertension, both of which are amenable to dietary sodium restriction. However, dietary change is widely known to be difficult to achieve and sustain. Controlling dietary sodium is particularly difficult for HD because many foods are naturally high in sodium, and most prepared/prepackaged foods have significant amounts of sodium added to enhance taste and shelf-life. Research on behavioral methods that are effective in reducing dietary sodium intake in HD is very limited. The purpose of this study is to test, in a randomized clinical trial of 200 HD patients, a behavioral intervention, paired with personal digital assistant (PDA)-based dietary self-monitoring, to enhance adherence to dietary sodium restrictions. Specifically the investigators will: (a) Assess the impact of the intervention on average daily interdialytic weight gains (IDWG-A). (b) Examine the impact of the intervention on self-reported dietary sodium intake. The study hypotheses are that compared to the control group, the intervention group will: (1) demonstrate a statistically significant decline in IDWG-A over the 4-month intervention period, and (2) experience a greater decline in dietary sodium intake. Secondarily, the investigators will explore the impact of the intervention on: (a) pre-dialysis pulse pressure and mean arterial blood pressure, (b) hemodialysis dietary self-efficacy, and (c) intradialytic and postdialytic symptoms and general health-related quality of life. In addition, the investigators will characterize the barriers/facilitators to adherence to the HD dietary regimen and patient experience of the intervention through the use of qualitative methods. The intervention is based on Social Cognitive Theory (SCT). Self-monitoring within the context of the intervention is operationalized as PDA-based dietary recording using BalanceLog software. Participants randomized to the attention control will receive computerized dietary education. Attention control participants will be offered an abbreviated version of the intervention after the 4-month study period concludes. Differences in IDWG-A, pulse pressure, and mean arterial pressure will be examined using a random intercept linear regression modeling. Self-reported dietary sodium, self-efficacy, symptoms, and quality of life will be assessed at baseline, 6 weeks, and 4 month and differences will be examined using repeated measures modeling using GEE. Qualitative analysis of narrative data will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with end stage renal disease (ESRD) who are 18 years of age or older,
* Individuals who are literate,
* Community-dwelling adults who have been receiving maintenance dialysis for at least 3 months.

Exclusion Criteria:

* Individuals who cannot read or write,
* Individuals who do not speak English,
* Individuals who plan to move out of the area or change dialysis centers within the next 6 months,
* Individuals who have a life expectancy of less than 12 months,
* Individuals who are scheduled for a living donor transplant,
* Individuals who cannot see the PDA screen or use the stylus to make food selections from the PDA screen, or
* Individuals who live in an institutional setting in which they would have limited control over their dietary intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Sevick MA, Piraino BM, St-Jules DE, Hough LJ, Hanlon JT, Marcum ZA, Zickmund SL, Snetselaar LG, Steenkiste AR, Stone RA. No Difference in Average Interdialytic Weight Gain Observed in a Randomized Trial With a Technology-Supported Behavioral Intervention to Reduce Dietary Sodium Intake in Adults Undergoing Maintenance Hemodialysis in the United States: Primary Outcomes of the BalanceWise Study. J Ren Nutr. 2016 May;26(3):149-58. doi: 10.1053/j.jrn.2015.11.006. Epub 2016 Feb 9. PMID 26868602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 17 dialysis centers, from the 3 corporate chains, between September 2009 and September 2012. Of the 848 HD patients available, 257 were eligible, 191 consented, 185 provided baseline data, 179 were randomized, and 160 (89.4%) completed the final 16-week measurement assessment.
Groups:
- Intervention: Intervention participants continue to receive routine dialysis care, as well as a 16 week dietary counseling intervention based on Social Cognitive Theory. Dietary counseling is paired with Personal Digital Assistant-based dietary self-monitoring.
  Social Cognitive Theory based dietary counseling paired with personal digital assistant based self-monitoring: The intervention duration is 16 weeks. Intervention contacts are 2x/week for weeks 0-8, weekly for weeks 9-12, and every other week for weeks 13-16. Personal digital assistant dietary records are use to provide targetted counseling and engaged the participant in problem solving around dietary issues.
Period: Overall Study
Arm/Group | Intervention | Attention Control
Started | 93 | 86
Completed | 81 | 79
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Population: One attention control participant was hospitalized after enrollment and did not have a baseline data collection form.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Attention Control | Total
Number analyzed (Participants) | 93 | 85 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.5) | 60.8 (13.4) | 59.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 57 | 44 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 91 | 83 | 174
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 33 | 66
  White | 59 | 51 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 93 | 85 | 178
Etiology of ESRD [Count of Participants; unit: Participants] — Etiology of ESRD
  Participants
    Diabetes | 37 | 34 | 71
    Hypertension | 19 | 30 | 49
    Glomerular disease | 14 | 6 | 20
    Polycystic disease | 5 | 1 | 6
    Neoplasms/tumors | 9 | 4 | 13
    Other | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time Specific Interdialytic Weight Gain (Baseline)
Description: Average interdialytic weight gains (kg/day) were calculated for the 1 week period prior to baseline measurement.
Time Frame: Baseline
Population: Some participants have missing interdialytic weight gains due to missed hemodialysis treatments.
Measure: Mean (Standard Deviation); unit: kg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 88 | 80
kg/day | 1.2 (0.6) | 1.2 (0.5)

2. Primary Outcome: Time Specific Interdialytic Weight Gain (8 Weeks)
Description: Average interdialytic weight gains (kg/day) were calculated for the 1 week period prior to the 8-week measurement time point.
Time Frame: 8 weeks
Population: Some participants have missing interdialytic weight gains due to missed hemodialysis treatments.
Measure: Mean (Standard Deviation); unit: kg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 81 | 80
kg/day | 1.1 (0.6) | 1.2 (0.5)

3. Primary Outcome: Time Specific Interdialytic Weight Gain (12 Weeks)
Description: Average interdialytic weight gains (kg/day) were calculated for the 1 week period prior to the 12 week measurement time point.
Time Frame: 12 weeks
Population: Some participants have missing interdialytic weight gains due to missed hemodialysis treatments.
Measure: Mean (Standard Deviation); unit: kg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 80 | 79
kg/day | 1.2 (0.5) | 1.2 (0.5)

4. Primary Outcome: Time Specific Interdialytic Weight Gain (16 Weeks)
Description: Average interdialytic weight gains (kg/day) were calculated for the 1 week period prior to the 16 week measurement time point.
Time Frame: 16 weeks
Population: Some participants have missing interdialytic weight gains due to missed hemodialysis treatments.
Measure: Mean (Standard Deviation); unit: kg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 79
kg/day | 1.1 (0.6) | 1.2 (0.5)

5. Primary Outcome: Time Specific Dietary Sodium Intake (Baseline)
Description: Dietary sodium intake was assessed via three 24-hour dietary recalls, including 1 dialysis weekday, 1 non-dialysis weekday, and 1 non dialysis weekend day. Recalls were entered into Nutrition Data System for Research, with sodium intake averaged across the 3 recalls.
Time Frame: Baseline
Population: Some participants have missing sodium data due to missed dietary recalls.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 92 | 85
mg/day | 2555 (2090) | 2298 (957)

6. Primary Outcome: Time Specific Dietary Sodium Intake (8 Weeks)
Description: as for outcome 5
Time Frame: 8 weeks
Population: Some participants have missing sodium data due to missed dietary recalls.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 82 | 80
mg/day | 2316 (931) | 2573 (1139)

7. Primary Outcome: Time Specific Dietary Sodium Intake (16 Weeks)
Description: as for outcome 5
Time Frame: 16 weeks
Population: Some participants have missing sodium data due to missed dietary recalls.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 78
mg/day | 2371 (1483) | 2447 (1067)

8. Primary Outcome: Time Specific Change From Baseline in Dietary Sodium Intake (Baseline to 8 Weeks)
Description: Dietary sodium intake was assessed via three 24-hour dietary recalls, including 1 dialysis weekday, 1 non-dialysis weekday, and 1 non dialysis weekend day. Recalls were entered into Nutrition Data System for Research, with sodium intake averaged across the 3 recalls. The difference between measurement time points was determined.
Time Frame: Baseline to 8 weeks
Population: Some participants have missing sodium data due to missed dietary recalls.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 82 | 79
mg/day | -71 (1027) | 237 (991)

9. Primary Outcome: Time Specific Change From Baseline in Dietary Sodium Intake (Baseline to 16 Weeks)
Description: as for outcome 5
Time Frame: Baseline to 16 weeks
Population: Some participants have missing sodium data due to missed dietary recalls.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 77
mg/day | 59 (1483) | 131 (993)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study period (16 weeks).
Arm/Group | Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 1/93 | 2/86
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/86
Other Adverse Events (participants affected / at risk) | 0/93 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No